CLINICAL TRIAL: NCT00387790
Title: A Phase II Study of Motexafin-Gadolinium (NSC 695238, IND #55583) and Involved Field Radiation Therapy for Intrinsic Pontine Glioma of Childhood
Brief Title: Motexafin Gadolinium and Radiation Therapy in Treating Young Patients With Pontine Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01829; NCI-2012-01829 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000504107; COG-ACNS0222; ACNS0222 (Other: Children's Oncology Group); ACNS0222 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Results first posted 2014-02-05 (Estimated); Last update posted 2018-01-04 (Actual); Status verified 2017-12

CONDITIONS: Untreated Childhood Brain Stem Glioma
MeSH Terms: interventions — motexafin gadolinium; Radiotherapy, Conformal

ARMS (1):
- Arm I (Experimental): Patients receive motexafin gadolinium IV over 5-10 minutes once daily (prior to radiotherapy) 5 days a week for 6 weeks. Patients undergo focal cranial radiotherapy once daily 5 days a week for 6 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: motexafin gadolinium; Radiation: 3-dimensional conformal radiation therapy

INTERVENTIONS:
Drug: motexafin gadolinium — Given IV
  Other Names: gadolinium texaphyrin; Gd (III) Texaphryin; Gd-Tex; PCI-0120; Xcytrin
Radiation: 3-dimensional conformal radiation therapy — Undergo focal cranial radiotherapy
  Other Names: 3D conformal radiation therapy; 3D-CRT

SUMMARY:
This phase II trial is studying how well giving motexafin gadolinium together with radiation therapy works in treating young patients with pontine glioma. Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs, such as motexafin gadolinium, may make tumor cells more sensitive to radiation therapy. Giving motexafin gadolinium together with radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the effect of combining motexafin gadolinium with daily fractionated radiotherapy on 1-year event-free survival of pediatric patients with intrinsic pontine glioma (brain stem glioma).

SECONDARY OBJECTIVES:

I. Evaluate the effect of combining motexafin gadolinium with daily fractionated radiotherapy on 1-year overall survival of these patients.

II. Determine the toxicities of motexafin gadolinium in combination with radiotherapy in these patients.

OUTLINE: This is a multicenter study.

Patients receive motexafin gadolinium IV over 5-10 minutes once daily (prior to radiotherapy) 5 days a week for 6 weeks. Patients undergo focal cranial radiotherapy once daily 5 days a week for 6 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 3 years and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of intrinsic pontine glioma (brain stem glioma)

  * Clinical and radiographic (MRI) evidence of tumors that diffusely involve the brain stem (i.e., tumors that intrinsically [> 50% intra-axial] involve the pons or pons and medulla, pons and midbrain, or entire brain stem) allowed
  * Tumor may contiguously involve the thalamus or upper cervical cord
  * No more than 1 lesion/mass present at diagnosis
* Karnofsky performance status (PS) 60-100% (age > 16 years) OR Lansky PS 60-100% (age ≤ 16 years)
* Life expectancy ≥ 8 weeks
* Absolute neutrophil count ≥ 1,000/mm³
* Platelet count ≥ 100,000/mm³ (transfusion independent)
* Hemoglobin ≥ 10 g/dL (RBC transfusions allowed)
* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min OR creatinine normal for age/gender (0.4-1.7 mg/dL)
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT < 1.5 times ULN
* No known glucose-6-phosphate dehydrogenase (G6PD) deficiency

  * If family history suggestive of congenital hemolytic anemia, patient must be screened for G6PD with G6PD activity test prior to study entry
* No biliary obstruction
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior definitive therapy for this specific tumor
* No prior cranial radiotherapy
* Concurrent steroids and anticonvulsants allowed
* No concurrent proton therapy
* No concurrent intensity-modulated radiotherapy
* No concurrent anticancer chemotherapy
* No concurrent immunomodulating agents

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2007-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Bradley, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiation and Motexafin Gadolinium: Patients receive motexafin gadolinium IV over 5-10 minutes once daily (prior to radiotherapy) 5 days a week for 6 weeks. Patients undergo localized cranial radiotherapy once daily 5 days a week for 6 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.
  motexafin gadolinium: Given IV
  2-dimensional, 3-dimensional conformal, or intensity-modulated radiation therapy: Undergo localized cranial radiotherapy
Period: Overall Study
Arm/Group | Radiation and Motexafin Gadolinium
Started | 64
Completed | 50
Not Completed | 14
Not completed — Adverse Event | 5
Not completed — Lack of Efficacy | 2
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 3
Not completed — Ineligible for study | 2

BASELINE CHARACTERISTICS:
Arm/Group | Radiation and Motexafin Gadolinium
Number analyzed (Participants) | 64
Age, Continuous [Mean (Full Range); unit: years] — Patients found not to meet the eligibility requirements are excluded from the age baseline measure.
  years | 6 [1 to 17]
Sex: Female, Male [Count of Participants; unit: Participants] — Patients found not to meet the eligibility requirements were not included in the gender baseline measure.
  Participants
    Female | 34
    Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants] — Patients found not to meet the eligibility requirements are excluded from the race baseline measure.
  Participants
    American Indian or Alaska Native | 1
    Asian | 1
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 11
    White | 42
    More than one race | 0
    Unknown or Not Reported | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Patients found not to meet the eligibility requirements are excluded from the ethnicity baseline measure.
  Participants
    Hispanic or Latino | 7
    Not Hispanic or Latino | 52
    Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants] — Patients found not to meet the eligibility requirements are excluded from the region baseline measure.
  participants
    United States | 55
    Canada | 4
    Australia | 5

OUTCOME MEASURES:

1. Primary Outcome: One Year Event-free Survival (EFS)
Description: Percentage probability of being event-free at 1 year following enrollment.
Time Frame: One year after enrollment.
Population: Patients found not to meet the eligibility requirements are by group policy not followed for adverse events or outcome. The 2 patients who are ineligible were excluded from the Outcome Measure analysis.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Radiation and Motexafin Gadolinium
Number analyzed (Participants) | 62
percent probability | 20 [11 to 31]

2. Secondary Outcome: Overall Survival (OS)
Description: Percentage probability of being alive 1 year following enrollment.
Time Frame: One year after enrollment.
Population: Only eligible patients are included therefore two patients were excluded from analysis.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Radiation and Motexafin Gadolinium
Number analyzed (Participants) | 62
percent probability | 53 [39 to 64]

3. Secondary Outcome: The Number of Patients Who Experience at Least One Grade 3 or Higher CTC Version 4 Toxicity.
Description: Occurrence of serious toxicity defined as any grade 4 hematologic toxicity that persists for more than 7 days or requires platelet transfusions for a time period exceeding 7 days; any grade 3 or 4 non-hematologic toxicity with the exception of grade 3 nausea or vomiting which can be controlled within 7 days; grade 3 skin reaction; grade 3 transaminitis.
Time Frame: One cycle of chemotherapy and radiation therapy; expected to be 42 days of treatment.
Population: Only eligible patients are included in the analysis, therefore two patients were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation and Motexafin Gadolinium
Number analyzed (Participants) | 62
Participants | 31

ADVERSE EVENTS:
Description: Patients found not to meet the eligibility requirements are by group policy not followed for adverse events or outcome.
Arm/Group | Radiation and Motexafin Gadolinium
Serious Adverse Events (participants affected / at risk) | 11/62
Other Adverse Events (participants affected / at risk) | 29/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation and Motexafin Gadolinium (N=62)
Abducens nerve disorder (Nervous system disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Anaphylaxis (Immune system disorders) | 1
Ataxia (Nervous system disorders) | 1
Catheter related infection (Infections and infestations) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Extraocular muscle paresis (Eye disorders) | 1
Fever (General disorders) | 2
Hydrocephalus (Nervous system disorders) | 2
Hypotension (Vascular disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 2
Lymphocyte count decreased (Investigations) | 3
Pain (General disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Skin infection (Infections and infestations) | 1
Weight loss (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation and Motexafin Gadolinium (N=62)
Alanine aminotransferase increased (Investigations) | 6
Alkaline phosphatase increased (Investigations) | 1
Allergic reaction (Immune system disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Anaphylaxis (Immune system disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Apnea (Respiratory, thoracic and mediastinal disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Ataxia (Nervous system disorders) | 2
Bladder infection (Infections and infestations) | 1
Catheter related infection (Infections and infestations) | 1
Constipation (Gastrointestinal disorders) | 1
Cushingoid (Endocrine disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Dysphasia (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
External ear inflammation (Ear and labyrinth disorders) | 1
Facial nerve disorder (Nervous system disorders) | 1
Fatigue (General disorders) | 1
Glossopharyngeal nerve disorder (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Hydrocephalus (Nervous system disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hypertension (Vascular disorders) | 5
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Ileus (Gastrointestinal disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Irritability (General disorders) | 1
Lung infection (Infections and infestations) | 1
Lymphocyte count decreased (Investigations) | 7
Mucositis oral (Gastrointestinal disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neutrophil count decreased (Investigations) | 1
Otitis media (Infections and infestations) | 2
Pain (General disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2
Peripheral motor neuropathy (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Urine discoloration (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Weight gain (Investigations) | 3
White blood cell decreased (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less